CLINICAL TRIAL: NCT01508598
Title: Validation of Circulating Endothelial Cells and Microparticles in Youth
Status: Terminated | Type: Observational
Why Stopped: Not enough subjects enrolled to be able to analyze data.
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: 1108M02842
Record Dates: First submitted 2011-12-13; First posted 2012-01-12 (Estimated); Last update posted 2020-08-24 (Actual); Status verified 2020-08

CONDITIONS: Childhood Obesity; Bariatric Surgery Candidate
Keywords: Pediatric; Obesity; Bariatric surgery; Cardiovascular disease
MeSH Terms: conditions — Pediatric Obesity; Obesity; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — 10 mL of blood serum and 5 mL of blood plasma will be frozen in long-term storage for future study analyses and use. 8 mL of urine will be frozen in long-term storage for future study analyses and use.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Identification and validation of early chronic disease biomarkers in children is of paramount importance especially in the burgeoning arena of pediatric obesity research. Despite the presence of risk factors, few obese children develop overt cardiovascular disease (CVD) early in life. However, because CVD is a cumulative process occurring over time, identifying the earliest signs in order to intervene sooner may have a large impact on slowing its progression. Endothelial activation is one of the earliest detectable signs of the beginnings of CVD. However, accurately quantifying endothelial health in children has proven to be a major challenge. Direct measures of endothelial cell biology, such as circulating endothelial cells (CEC) and endothelial microparticles (EMP), have been extensively studied in adults and are associated with vascular diseases, CVD risk factors, and CVD events. Despite being well-validated in adults, CEC and EMP have not been formally evaluated as disease biomarkers in children and adolescents. Pediatric obesity is an ideal condition in which to validate CEC and EMP as disease biomarkers since adiposity in childhood is associated with CVD, type 2 diabetes mellitus, and premature death, later in life. The investigators primary focus in this study will be the evaluation of CEC and EMP as biomarkers of CVD risk and whether substantial changes in weight affect these biomarkers. The investigators propose to evaluate the change in levels of CEC and EMP in response to substantial weight loss in 32 adolescents with extreme obesity undergoing elective, clinically-indicated bariatric surgery.

DETAILED DESCRIPTION:
Identification and validation of early chronic disease biomarkers in children is of paramount importance especially in the burgeoning arena of pediatric obesity research. Despite the presence of risk factors, few obese children develop overt CVD early in life. However, the pathologic process of CVD begins in the first two decades of life, particularly in the presence of obesity. Because CVD is a cumulative process occurring over time, identifying the earliest signs in order to intervene sooner may have a large impact on slowing its progression. The challenge is identifying which obese youth have early vascular problems. Looking to the vascular endothelium for biomarkers of damage is a reasonable approach because of its prominent role in the origins of atherosclerosis. Endothelial activation is one of the earliest detectable signs of the beginnings of CVD and predicts subsequent atherosclerosis and future cardiovascular events. However, accurately quantifying endothelial health in children has proven to be a major challenge.

Brachial artery FMD is the most commonly-used method to quantify endothelial health in children. However, this technique is not widely applicable, even in the research setting, because it requires specialized equipment and a highly-trained technician. Moreover, results can be highly variable (especially across sites) due to operator dependence and intra-individual fluctuations in endothelial function. More direct measures of endothelial cell biology, such as CEC and EMP, may offer greater precision in characterizing the state of the endothelium and may be especially useful as risk-prediction biomarkers in youth since they are hallmarks of advanced endothelial cell distress, thereby identifying the highest-risk individuals. CEC and EMP have been extensively studied in adults and are associated with vascular diseases, CVD risk factors, and CVD events. Despite being well-validated in adults, CEC and EMP have not been formally evaluated as disease biomarkers in children and adolescents.

Pediatric obesity is an ideal condition in which to validate CEC and EMP as disease biomarkers since adiposity in childhood is associated with CVD, type 2 diabetes mellitus, and premature death later in life. In particular, extreme obesity is an especially high-risk condition associated with significant co-morbidities. Our primary focus in this study will be the evaluation of CEC and EMP as biomarkers of CVD risk, with a goal of validating CEC and EMP for use as vascular endpoints in pediatric research studies. We propose to evaluate the change in levels of CEC and EMP in response to substantial weight loss in adolescents with extreme obesity undergoing elective, clinically-indicated bariatric surgery.

Specific Aims:

1. Evaluate the effect of substantial weight loss on levels of CEC and EMP in adolescents with extreme obesity.

We hypothesize that levels of CEC and EMP will be significantly reduced following elective, clinically-indicated bariatric surgery in adolescents with extreme obesity. The magnitude of change in CEC and EMP levels will be correlated with the magnitude of weight loss and improvements in CVD risk factors and endothelial function following bariatric surgery.

We will enroll 32 children and adolescents (ages 8-17) who are scheduled for elective bariatric surgery. They will be evaluated prior to their surgery, six months after surgery and twelve months after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age 8-17 years old
* Currently scheduled for elective bariatric surgery

Exclusion Criteria:

* None

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Thirty-two children and adolescents, who are currently scheduled to undergo elective bariatric surgery.
Sampling Method: Non-Probability Sample
Enrollment: 390 (Actual)
Dates: Start 2012-02 (Actual); Primary Completion 2018-01-02 (Actual); Study Completion 2018-01-02 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Circulating Endothelial Cell (CEC) VCAM Expression at 12-months | Baseline and 12-months

SECONDARY OUTCOMES:
Change from Baseline in Circulating Endothelial Cell (CEC) Enumeration at 12-months | Baseline and 12 Months
Change from Baseline in Endothelial Microparticle (EMP) VCAM Expression at 12-months | Baseline and 12 Months
Change from Baseline in Endothelial Microparticle (EMP) Enumeration at 12-months | Baseline and 12 Months
Change from Baseline in Circulating Endothelial Cell (CEC) VCAM Expression at 6-months | Baseline and 6-Months
Change from Baseline in Circulating Endothelial Cell (CEC) Enumeration at 6-months | Baseline and 6-Months
Change from Baseline in Endothelial Microparticle (EMP) VCAM Expression at 6-months | Baseline and 6-Months
Change from Baseline in Endothelial Microparticle (EMP) Enumeration at 6-months | Baseline and 6-Months

CONTACTS AND LOCATIONS:
Overall Officials: Aaron S Kelly, Ph.D., Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

REFERENCES:
- [Derived] Fox CK, Northrop EF, Rudser KD, Ryder JR, Kelly AS, Bensignor MO, Bomberg EM, Bramante CT, Gross AC. Contribution of Hedonic Hunger and Binge Eating to Childhood Obesity. Child Obes. 2021 Jun;17(4):257-262. doi: 10.1089/chi.2020.0177. PMID 34061621
- [Derived] Fyfe-Johnson AL, Ryder JR, Alonso A, MacLehose RF, Rudser KD, Fox CK, Gross AC, Kelly AS. Ideal Cardiovascular Health and Adiposity: Implications in Youth. J Am Heart Assoc. 2018 Apr 13;7(8):e007467. doi: 10.1161/JAHA.117.007467. PMID 29654202